CLINICAL TRIAL: NCT05390580
Title: Neuromodulation Using Vagus Nerve Stimulation Following Ischemic Stroke as Therapeutic Adjunct
Acronym: NUVISTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Osvaldo J. Laurido-Soto, MD, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 202203086
Record Dates: First submitted 2022-05-05; First posted 2022-05-25 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; cytokines; large vessel occlusion; vagal nerve stimulator
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This is a randomized open-label, with blinded outcome pilot study to evaluate the effect on inflammatory laboratory values and explore clinical outcomes in patients who present with ischemic strokes due to large vessel occlusions and are treated with either current accepted management, or accepted management in addition to transcutaneous auricular vagal nerve stimulation.
Who Masked: Participant
Masking Description: Patients enrolled in the trial will be randomized to treatment with electrical stimulation to the auricular branch of the vagus nerve (intervention) or stimulation to the great auricular nerve (cervical nerve branch)(Sham) via an auricular, transcutaneous vagus nerve stimulator.. All patients will be fitted with the device, the investigators will attach adhesive contacts to the left ear. Patients are blinded to the intervention and study personnel will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator (Experimental): All patients will be fitted with the device, the investigator will attach adhesive contacts to the left ear. Stimulation sessions will occur for 20 minutes twice daily during the inpatient period, the investigator will stimulate the auricular branch of the vagus nerve. Patients' will be treated with the following parameters: frequency 20 Hz, pulse width 250 µm, and and a fixed intensity of 0.5 milliampere. The amplitude of stimulation may be reduced if a patient complains of discomfort at the site of stimulation.
  Interventions: Device: transcutaneous auricular vagal nerve stimulation
- Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham (Sham Comparator): All patients will be fitted with the device, the investigator will attach adhesive contacts to the left ear. Stimulation sessions will occur for 20 minutes twice daily during the inpatient period. Patients assigned to the controls arm will have electricity applied to the the great auricular nerve (cervical nerve branch), the lobule of the ear. The investigator will stimulate the lobule of the ear. Patients' will be treated with the following parameters: frequency 20 Hz, pulse width 250 µm, and and a fixed intensity of 0.5 milliampere. The amplitude of stimulation may be reduced if a patient complains of discomfort at the site of stimulation.
  Interventions: Device: Sham transcutaneous vagal nerve stimulation

INTERVENTIONS:
Device: transcutaneous auricular vagal nerve stimulation — Stimulus of the auricular branch of the vagal nerve with the transcutaneous auricular vagal nerve stimulation.
  Arms: Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator
Device: Sham transcutaneous vagal nerve stimulation — Patients assigned to the controls arm will have no electricity applied to the Auricular Branch of the Vagus Nerve. Stimulus will be provided to the lobule of the ear, which is not innervated by the Auricular Branch of the Vagus Nerve.
  Arms: Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham

SUMMARY:
This is a randomized open-label, with blinded outcome pilot study to evaluate the effect on inflammatory laboratory values and explore clinical outcomes in patients who present with ischemic strokes due to large vessel occlusions and are treated with either current accepted management, or accepted management in addition to transcutaneous auricular vagal nerve stimulation.

DETAILED DESCRIPTION:
Stroke is a leading cause of death and disability worldwide. Approximately 80% of strokes are caused by cerebral ischemia. Although stroke is the third leading cause of death after heart disease and cancer, it leads to permanent disabilities in 80% of survivors. Large vessel occlusions (LVOs) account for up to 38% of acute ischemic strokes (AIS). LVOs represent a clinically significant subpopulation of cerebral ischemia due to their disproportionate morbidity and mortality without treatment. Up to 64% of patients without treatment of their LVO are dead or dependent at 3-6 months. Even after successful treatment (recanalization), infarcts can continue to increase in size, a process referred to as ischemia-reperfusion injury, for which even patients who are successfully treated in the acute setting can have poor outcomes. Highlighting the need for adjunct therapies to minimize ischemia progression for both post recanalized and unrecanalized patients. Neuroinflammation has long been recognized as an important element of AIS pathology. In the acute phase of AIS, non-specific inflammatory markers such as C reactive protein, and classical pro-inflammatory cytokines are elevated and have been associated with aggravating brain injury.

An interesting avenue of research has now aimed to better understand, and eventually to target these inflammatory pathways to improve outcomes after AIS, with anti-inflammatory interventions trialed in humans. Although ongoing trials are occurring in AIS, the immunomodulation agents can be costly and have marked side effects, for which finding adjunct treatments that are easy to administer and with minimal side effects is of the utmost importance. Vagal nerve stimulation (VNS) has previously been established to have anti-inflammatory effects, and has been successfully demonstrated in other models of inflammatory conditions. Given these promising results in animal studies of AIS, and the established safety of the noninvasive transcutaneous auricular VNS (taVNS), the authors propose prospectively studying this non-morbid and safe intervention in our AIS patients due to LVO population at Barnes Jewish Hospital. Our central hypothesis is that implementing transcutaneous auricular vagal nerve stimulation (taVNS) in the acute period following an ischemic stroke due to a large vessel occlusion will attenuate the expected inflammatory response to the stroke and will curtail morbidity associated with inflammatory-mediated clinical endpoints (i.e., infarct progression). The investigators aim to determine if inflammatory markers in the blood are impacted in patients treated with noninvasive VNS, and as a secondary outcome track patient outcomes to better understand the impact on morbidity and mortality.

Patients enrolled in the trial will be randomized to treatment with electrical stimulation to the auricular branch of the vagus nerve (intervention) or stimulation to the great auricular nerve (cervical nerve branch)(Sham) via an auricular, transcutaneous vagus nerve stimulator. All patients will be fitted with the device, the investigators will attach adhesive contacts to the left ear. Stimulation sessions will occur for 20 minutes twice daily during the inpatient period. Patients will have electricity applied to the different nerves depending on the randomization, they will be treated with stimulation with the following parameters: frequency 20 Hz, pulse width 250 µm, and a fixed intensity of 0.5 milliampere. The amplitude of stimulation may be reduced if a patient complains of discomfort at the site of stimulation. The site of stimulation will be inspected daily before and after treatment to ensure there is no redness or irritation at the site. The investigators will obtain laboratory samples on admission, day 0, and every 1.5 days till day 5 or discharge (whichever occurs first) to assess the patients inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who present with acute ischemic strokes due to large vessel occlusions

Exclusion Criteria:

* <18 years old
* patients with presumed chronic large vessel occlusions
* NIHSS<6
* pre-morbid modified Rankin score (mRS) >2
* unable to initiate treatment under 36 hours from symptom discovery
* Chronic or severe infection
* life expectancy <3 months
* patients' undergoing active cancer or immunosuppressive/modulating therapy
* patients with sustained bradycardia on arrival with a heart rate <50 beats per minute.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laurido-Soto OJ, Tan G, Nielsen SS, Huguenard AL, Donovan KM, Xu I, Giles J, Dhar R, Adeoye O, Lee JM, Leuthardt E. Transcutaneous Auricular Vagus Nerve Stimulation Reduces Inflammatory Biomarkers after Large Vessel Occlusion Stroke: Results of a Prospective Randomized Open-Label Blinded Endpoint Trial. Transl Stroke Res. 2025 Dec 22;17(1):7. doi: 10.1007/s12975-025-01405-6. PMID 41428140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We randomized 40 participants; after applying all study eligibility criteria, we excluded five participants post-hoc and included 35 participants (17 treated, 18 sham)
Pre-assignment Details: Patients were randomized in a 1:1 ratio to either the stimulation or sham treatment group using SAS software (Version 9.4, SAS). A total of 80 patients were assigned to one of two groups based on a computer-generated randomization sequence using the RANUNI function with a fixed seed (43523483) to ensure reproducibility. The generated sequence was then sorted, and the first 40 patients were allocated to the stimulation group, while the remaining 40 were assigned to the sham group.
Groups:
- Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator: Patients enrolled in the trial were randomized to treatment with electrical stimulation via an auricular, transcutaneous vagus nerve stimulator. All patients are fitted with a portable Soterix© device, a transcutaneous electrical nerve stimulation unit, and are connected to two ear electrodes, applied to the left ear during treatment periods. For taVNS treatment, these ear electrodes are placed along the concha of the ear, while in sham treatments the electrodes are placed along the ear lobe to avoid stimulation of the auricular vagus nerve from tactile pressure alone in the absence of current. Stimulation parameters were selected based on prior studies that sought to maximize vagus somatosensory evoked potentials while avoiding perception of pain. Stimulation parameters will be 20 minutes duration, frequency of 20 Hz, 250µs pulse width, and an intensity of 0.5mA. Sham treatments will involve no electrical current to the auricular branch of the vagal nerve.
Period: Overall Study
Arm/Group | Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator | Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham
Started (We excluded five participants post-hoc due to not meeting our inclusion criteria on re-review.) | 20 | 20
Completed | 17 | 18
Not Completed | 3 | 2
Not completed — Physician Decision | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator | Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] — Age
  years | 68.1 (15.2) | 67.3 (12.5) | 67.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex
  Participants
    Female | 7 | 10 | 17
    Male | 10 | 8 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 6 | 8
    White | 15 | 12 | 27
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Modified rankin scale [Mean (Standard Deviation); unit: units on a scale] — 0-6 functional description of deficits/disability - 0 = normal, 6 = death Population: Mean value provided - calculated per group.
  units on a scale | 0.37 (0.32) | 0.28 (0.21) | 0.31 (0.68)
NIH Stroke Scale (NIHSS) [Mean (Standard Deviation); unit: units on a scale] — This is a clinical secondary exploratory endpoints. The NIH Stroke Scale (NIHSS) is a clinical tool used to assess stroke severity, the score ranges from 0 up to 42 (higher is more severe). It will be assessed daily by the investigators and at day 30 on follow up. The investigators will assess differences in NIHSS dependent of the intervention arm.
  units on a scale | 16.4 (6.6) | 15.7 (4.4) | 16 (5.5)
Reperfusion % [Mean (Standard Deviation); unit: Percentage] — Based on the Thrombolysis in Cerebral Infarction (TICI) score (A measurement of reperfusion) we determined the percentage reperfused. Reperfused = TICI score >= 2B
  Percentage | 76 (27.1) | 83.8 (31.5) | 80 (29.3)
Time from Last Known Normal to recanalization attempt [Mean (Standard Deviation); unit: hours] — Time to reperfusion/recanalization
  hours | 13.2 (11.1) | 9.8 (10.6) | 11.5 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Interleukin - 1b - Changes and Differences in the Levels
Description: The primary endpoint was change in inflammatory biomarkers from baseline to day 5, with samples obtained every 1.5 days. Interleukin-1β was the main analyte. Repeated measures were analyzed longitudinally using mixed-effects models (FDA guidance), specifying subject as a random effect to account for multiple observations. This approach accommodated irregular timing, missing data, and time-varying covariates. Models included treatment, time since last known normal, and their interaction to test group differences in biomarker trajectories. Time was modeled quadratically for cytokine and WBC outcomes to capture U-shaped temporal patterns. Interaction p-values assessed trajectory differences between taVNS and sham arms.
Time Frame: 5 days
Population: The unit of measure below is a measurement of the trajectory of the values of the outcome measurement of interest, effectively a reflection of the graph of the results, with the number reflecting the slope of the curve. These values were compared based on their treatment arm and differences amongst treatment groups with mixed effect models utilizing p-interact values that allow the distinguishing of outcome trajectories. (i.e. were they statistically significant).
Measure: Number (95% Confidence Interval); unit: percent change/day
Arm/Group | Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator | Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham
Number analyzed (Participants) | 17 | 18
percent change/day | -0.222 [-0.903 to 0.460] | 0.327 [-0.047 to 0.702]
Statistical Analysis 1: Comparison: Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator vs Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham; Repeated measures were analyzed with longitudinal mixed-effects models (FDA guidance), using subject as a random effect. This accounted for irregular timing, missing data, and time-varying covariates. Models included treatment, time since last known normal, and their interaction; quadratic time terms captured U-shaped cytokine/WBC patterns. Interaction p-values tested trajectory differences between taVNS and sham; Test type: Superiority; p = 0.24, Mixed Models Analysis

2. Primary Outcome: Interleukin - 6 - Changes and Differences in the Levels
Description: The primary endpoint was change in inflammatory biomarkers from baseline to day 5, with samples obtained every 1.5 days. Interleukin-6 was the main analyte. Repeated measures were analyzed longitudinally using mixed-effects models (FDA guidance), specifying subject as a random effect to account for multiple observations. This approach accommodated irregular timing, missing data, and time-varying covariates. Models included treatment, time since last known normal, and their interaction to test group differences in biomarker trajectories. Time was modeled quadratically for cytokine and WBC outcomes to capture U-shaped temporal patterns. Interaction p-values assessed trajectory differences between taVNS and sham arms.
Time Frame: 5 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent change/day
Arm/Group | Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator | Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham
Number analyzed (Participants) | 17 | 18
percent change/day | -4.099 [-7.655 to -0.543] | 4.323 [2.369 to 6.277]
Statistical Analysis 1: Comparison: Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator vs Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0001, Mixed Models Analysis

3. Primary Outcome: Tumor Necrosis Factor Alpha - Changes and Differences in the Levels
Description: The primary endpoint was change in inflammatory biomarkers from baseline to day 5, with samples obtained every 1.5 days. Tumor necrosis factor was the main analyte. Repeated measures were analyzed longitudinally using mixed-effects models (FDA guidance), specifying subject as a random effect to account for multiple observations. This approach accommodated irregular timing, missing data, and time-varying covariates. Models included treatment, time since last known normal, and their interaction to test group differences in biomarker trajectories. Time was modeled quadratically for cytokine and WBC outcomes to capture U-shaped temporal patterns. Interaction p-values assessed trajectory differences between taVNS and sham arms.
Time Frame: 5 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent change/day
Arm/Group | Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator | Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham
Number analyzed (Participants) | 17 | 18
percent change/day | -0.244 [-0.545 to 0.058] | -0.120 [-0.597 to 0.357]
Statistical Analysis 1: Comparison: Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator vs Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.26, Mixed Models Analysis

4. Primary Outcome: White Blood Cell Total Count - Changes and Differences in the Levels
Description: The primary endpoint was change in inflammatory biomarkers from baseline to day 5, with samples obtained every 1.5 days. WBC count was the main analyte. Repeated measures were analyzed longitudinally using mixed-effects models (FDA guidance), specifying subject as a random effect to account for multiple observations. This approach accommodated irregular timing, missing data, and time-varying covariates. Models included treatment, time since last known normal, and their interaction to test group differences in biomarker trajectories. Time was modeled quadratically for cytokine and WBC outcomes to capture U-shaped temporal patterns. Interaction p-values assessed trajectory differences between taVNS and sham arms.
Time Frame: 5 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent change/day
Arm/Group | Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator | Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham
Number analyzed (Participants) | 17 | 18
percent change/day | -0.914 [-1.687 to -0.141] | -0.050 [-0.455 to 0.356]
Statistical Analysis 1: Comparison: Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator vs Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.14, Mixed Models Analysis

5. Primary Outcome: Neutrophil to Lymphocyte Ratio - Changes and Differences in the Levels
Description: The primary endpoint was change in inflammatory biomarkers from baseline to day 5, with samples obtained every 1.5 days. neutrophil to lymphocyte ratio based on blood samples was the main result of interestse. Repeated measures were planned to be analyzed longitudinally using mixed-effects models (FDA guidance), specifying subject as a random effect to account for multiple observations. This approach accommodated irregular timing, missing data, and time-varying covariates. Models included treatment, time since last known normal, and their interaction to test group differences in biomarker trajectories.
Time Frame: 5 days
Population: We were unable to analyze this outcome due to no patient (0/35) in the trial obtaining a repeat Complete blood count (CBC) with differential within the 5 days post baseline/recruitment. 15% patients underwent a repeat CBC with differential after day 7, outside of our analysis window.
Measure: Number; unit: ratio
Arm/Group | Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator | Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham
Number analyzed (Participants) | 17 | 18
ratio | NA — We were unable to analyze this outcome due to a lack of CBC with differentials as standard of care, 0% of our patients underwent follow up CBC with differential in the initial 5 days. | NA — We were unable to analyze this outcome due to a lack of CBC with differentials as standard of care, 0% of our patients underwent follow up CBC with differential in the initial 5 days.

6. Secondary Outcome: Change in NIH Stroke Scale (NIHSS)
Description: The secondary endpoint was change in NIHSS from baseline to discharge (~ day 5) and 30 days. Change in the NIHSS stroke scale number (0-42 and a measure of severity) was the outcome of interest. Repeated measures were analyzed longitudinally using mixed-effects models (FDA guidance), specifying subject as a random effect to account for multiple observations. This approach accommodated irregular timing, missing data, and time-varying covariates. Models included treatment, time since last known normal, and their interaction to test group differences in biomarker trajectories. Time was modeled quadratically for cytokine and WBC outcomes to capture U-shaped temporal patterns. Interaction p-values assessed trajectory differences between taVNS and sham arms and linearly for in-hospital NIHSS scores based on panel data plots. Interaction terms were utilized to delineate differences amongst trajectories of the outcome of interest.
Time Frame: 30 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: score change/day
Arm/Group | Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator | Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham
Number analyzed (Participants) | 17 | 18
score change/day | -1.613 [-2.576 to -0.651] | -1.562 [-5.25 to -0.978]
Statistical Analysis 1: Comparison: Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator vs Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham; Repeated measures were analyzed with longitudinal mixed-effects models (FDA guidance), using subject as a random effect. This accounted for irregular timing, missing data, and time-varying covariates. Models included treatment, time since last known normal, and their interaction; linearly for in-hospital NIHSS scores based on panel data plots. Interaction terms were utilized to delineate differences amongst trajectories of the outcome of interest; Test type: Superiority; p = 0.69, Mixed Models Analysis

7. Secondary Outcome: Modified Ranking Scale (mRS)
Description: This is a clinical secondary exploratory endpoints. The Modified Ranking Scale (mRS) is a clinical tool used to assess functional status after suffering a stroke. It ranges from 0 up to 6. It was assessed at day 90. The investigators will assess differences in mRS dependent of the intervention arm.
  0 = no symptoms at all
  1. = No significant disability despite symptoms; able to carry out all usual duties and activities
  2. = Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance.
  3. = Moderate disability; requiring some help, but able to walk without assistance.
  4. = Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. = Severe disability; bedridden, incontinent and requiring constant nursing care and attention.
  6. = Dead
Time Frame: 90 days
Population: There were three patients lost to follow up in the treatment group and one patient lost to follow up in the sham group, for which we utilized the 14 patients in the treatment group and the 17 patients left for the analyses, as we were not able to have data for the full recruited patients for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator | Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham
Number analyzed (Participants) | 14 | 17
score on a scale | 3.27 (2.15) | 2.78 (2.07)
Statistical Analysis 1: Comparison: Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator vs Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham; Estimated using a mixed model that includes a random effect for person, based on actual day of the mRS, 90 day assessment. Restricted to participants who survived to an mRS assessment for day 90 , leaving 14 participants (28 mRS scores) in the treatment group and 17 participants (34 mRS scores) in the sham group; Test type: Superiority; p = 0.48, Mixed Models Analysis

8. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0 - Hypotension (C143352)
Description: The investigator will monitor the patient's blood pressure (millimeters of mercury - mmHg) before, during, and after the transauricular vagal nerve stimulation or sham. If hypotension occurs (systolic blood pressure less than 80 mmHg or mean arterial pressure <60 mmHg) , the investigator will document it and assigned the appropriate grade from 1-5 based on the CTCAE.
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator | Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham
Number analyzed (Participants) | 17 | 18
Participants | 0 | 2
Statistical Analysis 1: Comparison: Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator vs Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham; To assess our dichotomous safety endpoints, we used logistic regression models constructed to assess differences in hypotension; Test type: Equivalence — Here we were testing if there were any safety differences based on treatment. This was a pilot exploratory trial, for which we may be underpowered; p = 0.49, Regression, Logistic

9. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0 - Sinus Bradycardia (C54940)
Description: The investigator will monitor the patient's heart rate (beat per minute) before, during, and after the transauricular vagal nerve stimulation or sham. If Sinus Bradycardia (C54940) occurs (heart rate less than 60 beats per minute), the investigator will document it and assigned the appropriate grade from 1-5 based on the CTCAE.
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator | Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham
Number analyzed (Participants) | 17 | 18
Participants | 2 | 4
Statistical Analysis 1: Comparison: Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator vs Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham; To assess our dichotomous safety endpoints, we used logistic regression models constructed to assess differences in bradycardia; Test type: Equivalence — [test comment as in outcome 8, analysis 1]; p = 0.66, Regression, Logistic

ADVERSE EVENTS:
Time Frame: enrollment until end of follow-up (up to 105 days).
Description: All adverse events were address in real time while the patients were inpatient and later at follow up.
Arm/Group | Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator | Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham
All-Cause Mortality (participants affected / at risk) | 3/17 | 2/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 2/17 | 6/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stimulation with Transcutaneous Auricular Vagal Nerve Stimulator (N=17) | Control - Transcutaneous Auricular Vagal Nerve Stimulator - Sham (N=18)
The above patient events were bradycardia and hypotension, none were serious. (Cardiac disorders) | 2 (2) | 6 (6) — Determined by reviewing the vital signs and talking to the ICU or primary teams.

LIMITATIONS AND CAVEATS:
1) the small sample size introduces the possibility that our findings may be subject to chance variation. 2) not powered to detect clinical differences. 3) fundamental questions remain about optimal therapeutic parameters, including stimulation settings, treatment duration, and most relevant physiologic and biomarker endpoints when utilizing taVNS. Please see manuscript attached for further details.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT05390580/Prot_SAP_ICF_001.pdf